CLINICAL TRIAL: NCT02614755
Title: An Observational Study of Lumosity in Seniors
Status: Completed | Type: Observational
Sponsor: Lumos Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LL004
Record Dates: First submitted 2015-11-18; First posted 2015-11-25 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
Keywords: Older Adults Volunteers; Seniors; Brain Performance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this observational study is to determine performance characteristics and usability of Lumosity and the Brain Performance Test in a group of older adult volunteers.

DETAILED DESCRIPTION:
Approximately 200 prospective users currently will be provided free 6-month premium access Lumosity accounts. Participants will be provided with an account activation code and instructed on how to sign up for Lumosity with their email address. They will be subject to the Lumosity Terms of Service and follow the typical user experience. Upon creating an account, users would be asked to complete a short demographic survey that includes questions on gender, education, occupation, years since retirement, health, computer familiarity, and perceptions of brain training.

Those who sign up will have immediate access to the Lumosity training system and the entire suite of Lumosity games. In addition, they will be invited, via email, to take the Brain Performance Test one week after the initial sign-up and then again 12 weeks later. Approximately every 8 weeks, users will be asked to complete a short questionnaire about their experience with Lumosity. This questionnaire will be accessed via email. Participants will be asked to train 5 days a week for 20-30 minutes per day, but are free to play as much or a little as they choose. Community associates at the sites will be encouraged to host group training sessions, giving the seniors a chance to gather and complete their training together, share their experiences, and get any help they may need. In addition, sites will have the option of hosting 1-2 focus groups with participants and researchers from Lumos Labs. The focus groups will be an opportunity to give and receive direct feedback about Lumosity, and get any questions answered by the researchers.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria:

1. 55 years of age or older
2. English-speaker
3. Cognitively stable (i.e., without a known diagnosis that may affect cognitive abilities)
4. Regular access to and ability to use a computer or mobile device with Internet connectivity.

Exclusion Criteria:

1. Under 55 years of age
2. Have a current diagnosed cognitive or neuropsychological condition
3. Are taking medication that may impede cognitive functioning
4. Anticipate a dosage change in medication that may affect cognitive functioning during the course of the study (24 weeks)
5. Have other conditions or problems that may preclude regular computer usage

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants must be cognitively stable older adult volunteers(over 55 years of age)
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-11; Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Usability - as measured by self-report feedback surveys | Change from Baseline - collected at baseline, 3 months and 6 months
  Using self-report surveys administered to participants at baseline, 3 months and 6 months, investigators will calculate a usability score of Lumosity.

SECONDARY OUTCOMES:
User Engagement - as measured by number of unique days played | 6 months
  Calculating the number of unique days played will allow us to estimate the engagement level of study participants.
Change from baseline on the Lumosity Performance Index (LPI) | Change from Baseline - collected at baseline and 6 months
  To evaluate the Lumosity Performance Index (LPI) results in a group of seniors
Change from baseline on the Brain Performance Test (BPT) | Change from Baseline - collected at baseline, 3 months and 6 months
  To evaluate the Brain Performance Test (BPT) results in a group of seniors

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Morrison, PhD, Principal Investigator — Lumos Labs
Locations (1):
- Lumos Labs, Inc., San Francisco, California, United States